CLINICAL TRIAL: NCT01222897
Title: An Open Label, Balanced, Randomized, Two-treatment, Two-period, Two-sequence, Single-dose, Crossover, Bioequivalence Study Comparing Valacyclovir Hydrochloride Tablets 1 Gram of Ohm Laboratories Inc. (A Subsidiary of Ranbaxy Pharmaceuticals Inc., USA) With VALTREX® Caplets 1 Gram (Containing Valacyclovir Hydrochloride 1 Gram) of GlaxoSmithKline in Healthy, Adult, Male, Human Subjects Under Fed Condition.
Brief Title: A Relative Bioavailability Study of Valacyclovir Hydrochloride Tablets 1gm Under Fed Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 216_VALAC_09
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2010-10

CONDITIONS: Healthy
Keywords: Valacyclovir hydrochloride fed study
MeSH Terms: interventions — Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Valacyclovir hydrochloride tablets 1 gm of OHM Laboratories Inc. (a subsidiary of Ranbaxy Pharmaceuticals Inc.)
  Interventions: Drug: Valacyclovir hydrochloride
- Reference (Active Comparator): VALTREX® (valacyclovir HCl) caplets 1 gm of GlaxoSmithKline Research Triangle Park, NC 27709
  Interventions: Drug: Valacyclovir hydrochloride

INTERVENTIONS:
Drug: Valacyclovir hydrochloride

SUMMARY:
The study was conducted as an open-label, balanced, randomized, two-treatment, two-period, two-sequence, single-dose, crossover, bioequivalence study comparing Valacyclovir hydrochloride tablets 1 gram manufactured by OHM Laboratories Inc. NJ 08901 with VALTREX® caplets 1 gram manufactured by GlaxoSmithKline, Research Triangle Park, NC 27709 in healthy, adult, male, human subjects under fed condition.

DETAILED DESCRIPTION:
Following an overnight fast of at least 10 hour, a high-fat high-calorie breakfast was served to the study subjects. Thirty minutes after start of this breakfast, a single oral dose of Valacyclovir hydrochloride 1 gram of either test or reference investigational product was administered during each period of the study (on day 01 and 04), along with 240 mL of drinking water at ambient temperature under low light condition and under supervision of trained study personnel. Both test and reference products were administered to all the study subjects, one in each period (except subject number 14 who dropped out from the study and subject number 37 who was withdrawn from the study).

During the course of the study, safety parameters assessed were vital signs, clinical examination, medical history and clinical laboratory safety tests (hematology, biochemical parameters, serology and urine analysis) at baseline. Adverse event monitoring was done throughout the study. Laboratory parameters of hematology and biochemistry (except blood glucose and cholesterol) were repeated at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Were in the age range of 18-45 years.
* Were neither overweight nor underweight for his height as per the Life Insurance Corporation of India height/weight chart for non-medical cases.
* Had voluntarily given written informed consent to participate in this study.
* Were of normal health as determined by medical history and physical examination of the subjects performed within 21 days prior to the commencement of the study.
* Had non-vegetarian dietary habit.

There were no deviations in this regard.

Exclusion Criteria:

* History of known hypersensitivity to Valacyclovir, related drugs like Acyclovir or to any other drug.
* Any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
* Presence of disease markers of HIV 1 or 2, Hepatitis B or C viruses or syphilis infection.
* Presence of values which were out of acceptable limits for hemoglobin, total white blood cells count, differential WBC count or platelet count.
* Positive for urinary screen testing of drugs of abuse (opiates or cannabinoids).
* Presence of values which were out of acceptable limits for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol.
* Clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4/HPF), glucose (positive) or protein (positive).
* Clinically abnormal ECG or Chest X-ray.
* History of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or hematological disease, diabetes or glaucoma.
* Inability to communicate well (i.e. language problem, poor mental development, psychiatric illness or poor cerebral function) that might impair the ability to provide, written informed consent.
* Regular smokers who smoked more than 10 cigarettes daily or had difficulty abstaining from smoking for the duration of each study period.
* History of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or had difficulty in abstaining for the duration of each study period.
* Used any regular medication (OTC or prescription) with in 14 days or any drug metabolizing enzyme modifying medications within 30 days prior to Day 1 of this study.
* Participated in any clinical trial within 12 weeks preceding Day 1 of this study (except for the subjects who dropout/withdrawn from the previous study prior to period I dosing).
* Subjects who, through completion of this study, had donated and /or lost more than 350 ml of blood in the past 3 months other than study participation.

There were no deviations in this regard.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-05; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Bioequivalence evaluation of Valacyclovir Hydrochloride tablets 1gm under fasting conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Ranbaxy Clinical Pharmacology Unit, Ranbaxy Laboratories Limited, Noida, Uttar Pradesh, India

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html